CLINICAL TRIAL: NCT06631729
Title: Targeting Transdiagnostic Self-regulatory Factors and Eating Disorder Pathology Among Adults With BInge-spectrum Eating disOrders: A mHEALTH Interoceptive Exposure Intervention (the Bio-HEALTH Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: the Bio-HEALTH Study
Record Dates: First submitted 2024-09-29; First posted 2024-10-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): randomized to HRV bio
  Interventions: Behavioral: HRV-bio
- Group 2 (Experimental): Randomized to ED-JITAI treatment
  Interventions: Behavioral: ED-JITAI

INTERVENTIONS:
Behavioral: HRV-bio — participants will complete a HRV biofeedback task via the Elite HRV app. In this intervention, participants will learn how to use their HRV data that they will see in real-time via the Elite HRV app to improve their HRV by engaging in an app-guided diaphragmatic breathing exercise. They will complete this exercise twice daily (morning, night).
  Arms: Group 1
Behavioral: ED-JITAI — participants will be prompted to complete focused, guided body scan tasks that will be sent to them via the MindLogger app. These guided tasks will be sent to them in the form of 1 of 3 brief (3-5 minute) videos via the MindLogger app. The body scans will be designed to promote participants' connection with, vs.
  distancing/distraction from, feared ED sensations (e.g., hunger, satiety, bloating).
  Participants will receive prompts to complete the body scans at times when they report via EMA that they are experiencing worse interoception than usual. "Worse interoception than usual" will be defined as participants' EMA-reported interoception scores during the intervention period that fall 1 SD or more above their baseline EMA-reported interoception levels.
  Arms: Group 2

SUMMARY:
The present study will be fully remote (virtual) and include observational design features (assessments) plus a clinical trial. All assessments will be completed using HIPAA-approved platforms (e.g., Qualtrics, MindLogger EMA platform). After screening via Qualtrics to determine eligibility (described below), participants will complete a cross-sectional survey via Qualtrics, followed by a baseline EMA period. During the baseline EMA period, participants will receive brief (3-5 minutes) surveys on their mobile devices 6 times per day for 7-days via the MindLogger app. During the baseline EMA period, participants will also be asked to wear non-invasive chest-worn Holter monitors (Polar H10 Holter monitors) that will capture their heartrate variability data.

They will then complete the 4-week intervention (HRV bio or ED-JITAI treatment arms; see below), followed by a post-intervention 7-day EMA assessment period while they also wear the Holter monitors. Recruitment is expected to last for 1.5 years. In HRV-bio, participants will also complete a HRV biofeedback task via the Elite HRV app. In this intervention, participants will learn how to use their HRV data that they will see in real-time via the Elite HRV app to improve their HRV by engaging in an app-guided diaphragmatic breathing exercise. They will complete this exercise twice daily (morning, night). In ED-JITAI, participants will be prompted to complete focused, guided body scan tasks that will be sent to them via the MindLogger app. These guided tasks will be sent to them in the form of 1 of 3 brief (3-5 minute) videos via the MindLogger app. The body scans will be designed to promote participants' connection with, vs.

distancing/distraction from, feared ED sensations (e.g., hunger, satiety, bloating).

Participants will receive prompts to complete the body scans at times when they report via EMA that they are experiencing worse interoception than usual. "Worse interoception than usual" will be defined as participants' EMA-reported interoception scores during the intervention period that fall 1 SD or more above their baseline EMA-reported interoception levels.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-64;
* no changes to ED treatment in the past 4-weeks;
* agree not to access other eating disorder treatments throughout the studies (unless warranted by a worsening of participants' symptoms during the study period; see Monitoring Participant Safety for more information);
* no bariatric surgery (prior or planned during the study period);
* no pregnancy or lactation (current or planned during the study);
* own an Apple or Android-brand iOS smartphone (which is required for compatibility with the apps used in this study;
* reside in the continental U.S.;
* meet Diagnostic and Statistical Manual of Mental Disorders-5-TR (DSM-5-TR) criteria for binge eating disorder (BED) or bulimia nervosa (BN), both of which include objective binge eating (i.e., consuming a larger amount of food than most people would eat in a similar period of time under similar circumstances with loss of control over eating during the episode) ≥1x/week over the past 3 months (APA, 2022). Single-item questions will determine eligibility via criteria 1-7. Criterion 8 for will be determined via the Eating Disorder Diagnostic Scale for the DSM-5 (EDDS-5; Stice et al., 2000, 2004), which has exhibited good sensitivity (.88), specificity (.98), and positive predictive power (.74) for detecting EDs among community samples (Stice et al., 2000, 2004).

Exclusion Criteria:

* not between the ages of 18 and 64;
* had changes to ED treatment in the past 4 weeks;
* plan to access other eating disorder treatments throughout the study;
* received or are planning to undergo bariatric surgery during the study period;
* currently pregnant or lactating, or planning to become pregnant or lactate during the study period;
* no Apple or Android-brand iOS smartphone;
* do not live in the continental U.S.;
* do not currently experience BN or BED.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Momentary binge eating | baseline, 5 weeks
  "Momentary binge eating" is operationalized as an eating episode in which participants report that they consumed an unusually large amount of food, given the circumstances, while also experiencing a loss of control over their eating at that time. This construct will be assessed at the momentary (or state) level of analysis using ecological momentary assessment.
Momentary purging behaviors | baseline, 5 weeks
  "Momentary purging behaviors" include the following behaviors that individuals may engage in at a given moment as maladaptive attempts of preventing weight gain or losing weight: self-induced vomiting; maladaptive use of laxatives; maladaptive use of diuretics; fasting (e.g., no food for >8 hours, skipping meals); excessive exercise. These behaviors will be assessed at the momentary (or state) level of analysis using ecological momentary assessment.
Heartrate variability | baseline, 5 weeks
  Heartrate variability is a generalized neurobiological indicator of interoception (the ability to sense and connect with one's internal bodily sensations) and autonomic nervous system functioning. It will be assessed using Holter monitors and smartwatches that capture fluctuations in the time intervals between adjacent heartbeats.
Momentary self-reported interoceptive sensibility | baseline, 5 weeks
  "Momentary self-reported interoceptive sensibility" is operationalized as individuals' subjective (selfreported) perceptions of their ability to sense and connect with their internal body sensations at a given moment, such as hunger, satiety, heartbeat, pain, bloating, etc. This construct will be assessed at the momentary (or state) level of analysis using ecological momentary assessment.
Treatment Compliance | baseline, 5 weeks
  For participants in the HRV-bio intervention arm, treatment compliance is operationalized as the number of HRV-biofeedback tasks that participants complete during the 4-week intervention period ÷ the total possible number of HRV-biofeedback tasks. For participants in the ED-JITAI intervention arm, treatment compliance is operationalized as the number of app-prompted focused body scans that participants complete during the 4-week intervention period ÷ the total possible number of focused body scans that they are prompted to complete. The total possible number of focused body scans will differ for each participant, as they will only receive prompts to complete these scans when they report via ecological momentary assessment that they are experiencing worse interoception than usual (with "usual" determined based on their personal mean interoception values that will be obtained during the pre-treatment ecological momentary assessment period).
Attrition | baseline, 5 weeks
  Attrition is operationalized as the total number of participants who stop participating in the 4-week intervention prematurely, as evidenced by a complete cessation of engaging in the intervention tasks (HRV-biofeedback task or focused body scan prompts), or who are otherwise lost to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Peterson, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT06631729/ICF_000.pdf